CLINICAL TRIAL: NCT05669482
Title: A Phase 1b/2a Study of Gemcitabine and Nab-paclitaxel in Combination With Avutometinib (VS-6766) and Defactinib in Patients With Previously Untreated Metastatic Adenocarcinoma of the Pancreas
Brief Title: Study of Avutometinib (VS-6766) +Defactinib With Gemcitabine and Nab-paclitaxel in Patients With Pancreatic Cancer
Acronym: RAMP205
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-205
Record Dates: First submitted 2022-12-06; First posted 2022-12-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: KRAS Activating Mutation; Metastatic Cancer; Pancreas Cancer; Neoplasms Pancreatic; Malignant Neoplasm of Pancreas
Keywords: avutometinib (VS-6766); Metastatic Cancer; KRAS Mutation; Pancreatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms | interventions — defactinib; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemcitabine + nab-paclitaxel + avutometinib (VS-6766) + defactinib (Experimental): To determine the recommended phase 2 dose (RP2D) for gemcitabine Gemcitabine + nab-paclitaxel + avutometinib (VS-6766) + defactinib in patients with untreated metastatic PDAC.
  Interventions: Drug: avutometinib (VS-6766) and defactinib in combination with gemcitabine and nab-paclitaxel
- Gemcitabine + nab-paclitaxel + avutometinib (VS-6766) + defactinib RP2D (Experimental): To determine the efficacy of the RP2D identified in Part A in untreated metastatic PDAC patients
  Interventions: Drug: avutometinib (VS-6766) and defactinib in combination with gemcitabine and nab-paclitaxel

INTERVENTIONS:
Drug: avutometinib (VS-6766) and defactinib in combination with gemcitabine and nab-paclitaxel — The RP2D of avutometinib (VS-6766) and defactinib in combination with gemcitabine and nab-paclitaxel determined in Part A will be used in Part B dose expansion.
  Other Names: Gemzar; Abraxane

SUMMARY:
This study will assess the safety and efficacy of avutometinib (VS-6766) and defactinib in combination with gemcitabine and nab-paclitaxel in patients with Pancreatic Ductal Adenocarcinoma (PDAC) who have been previously untreated.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open-label Phase 1/2 study designed to evaluate safety, tolerability and efficacy of avutometinib (VS-6766) and defactinib in combination with gemcitabine and nab-paclitaxel in patients previously untreated metastatic Pancreatic Ductal Adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age
* Histologic or cytologic evidence of metastatic pancreatic ductal adenocarcinoma.
* An Eastern Cooperative Group (ECOG) performance status ≤ 1
* Measurable disease according to RECIST 1.1
* Adequate organ function
* Adequate cardiac function
* Agreement to use highly effective method of contraceptive

Exclusion Criteria:

* Patients with pancreatic neuroendocrine tumors
* Prior or concomitant treatment for metastatic pancreatic ductal adenocarcinoma
* Prior treatment with inhibitors of the RAS /MAPK pathway [e.g. MEK inhibitors] or inhibitors of FAK
* History of prior malignancy, with the exception of curatively treated malignancies
* Major surgery within 4 weeks (excluding placement of vascular access)
* Concurrent heart disease or severe obstructive pulmonary disease
* Concurrent ocular disorders
* Active skin disorder that has required systemic therapy within the past 1 year
* Patients with interstitial lung disease or pulmonary fibrosis or severe lung disease, pulmonary edema, and adult respiratory distress syndrome
* Known SARS-Cov2 infection ≤28 days prior to first dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Part A: To determine RP2D for avutometinib (VS-6766) and defactinib in combination gemcitabine and nab-paclitaxel | 28 days
  Assessment of Dose-limiting toxicities (DLTs)
To determine the efficacy of the RP2D identified in Part A | 6 months
  Confirmed overall response rate (ORR) (partial response [PR] + complete response [CR] defined according to Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1])

SECONDARY OUTCOMES:
Duration of Response (DOR) | 24 months
  Time of first response to PD as assessed per RECIST 1.1
Disease Control Rate (DCR) | 24 months
  CR + PR + SD as assessed per RECIST 1.1
Progression Free Survival (PFS) | 24 months
  From the time of first dose of study intervention to PD as assessed per RECIST 1.1 or death from any cause
Overall Survival (OS) | Up to 5 years
  From the time of first dose of study intervention to PD as assessed per RECIST 1.1 or death from any cause
Plasma Pharmacokinetics (PK) of avutometinib (VS-6766) and Defactinib and relevant metabolites, Tmax | 10 weeks
  Time to Maximum concentration (Tmax)
Plasma Pharmacokinetics (PK) of avutometinib (VS-6766) and Defactinib and relevant metabolites, AUC | 10 Weeks
  Area under plasma Concentration (AUC) 0 to t
Plasma Pharmacokinetics (PK) of avutometinib (VS-6766) and Defactinib and relevant metabolites, Half-life | 10 weeks
  concentration Half-life (T1/2)
Frequency and severity adverse events (AEs) and Serious Adverse Events (SAEs) | 24 months
  Count of AE and SAEs by grade, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale
Number of abnormal laboratory values | 24 months
  Count of abnormal laboratory values by grade

CONTACTS AND LOCATIONS:
Overall Officials: MD Verastem, Study Director — Verastem, Inc.
Locations (12):
- United States (12):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - New York Presbyterian/Weill-Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No